CLINICAL TRIAL: NCT00581607
Title: Double Blind, Randomized Trial of Bosentan for Sarcoidosis Associated Pulmonary Hypertension
Acronym: BOSAPAH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOSAPAH-1; 7-3-22-1
Record Dates: First submitted 2007-12-26; First posted 2007-12-27 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoidosis; Pulmonary Arterial Hypertension
Keywords: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis; Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan for 16 weeks (Active Comparator): Active drug
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): Placebo for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — 62.5 mg bid for 4 weeks, then 125 mg bid
  Other Names: Tracleer
  Arms: Bosentan for 16 weeks
Drug: Placebo — Placebo twice a day
  Arms: Placebo
Drug: Bosentan — drug given for 16 weeks
  Other Names: tracleer
  Arms: Bosentan for 16 weeks
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Patients with advanced sarcoidosis often develop pulmonary hypertension. Pulmonary hypertension is a condition where the right side of the heart has to push the blood though the lungs at a higher pressure than normal. Since this pressure is higher, it is harder for the heart to pump the blood through the lungs to the left side of the body. If the blood can not get through the lungs, it can not get pumped through the rest of the body. This leads to weakness and shortness of breath. This type of hypertension does not usually respond to regular blood pressure medicines. The purpose of this study is to determine if bosentan (Tracleer) will help sarcoidosis associated pulmonary hypertension.

DETAILED DESCRIPTION:
Patients will be randomized in 2:1 manner to receive either bosentan or placebo for 16 weeks. After 16 weeks, there will be an additional 32 weeks of an open label extension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known sarcoidosis 21.
* Age 18 or greater
* Patients with documented pulmonary hypertension with a PA mean > 25 mm Hg as measured by cardiac catheterization within six months of entry into the study. Pulmonary artery occluding pressure and or left ventricular end diastolic pressure must be less than 15 mm Hg.
* Patients with WHO class II or III
* Six minute walk distance of between 100 to 500 meters
* Patients on stable immunotherapy for their sarcoidosis, including prednisone, methotrexate, azathioprine, hydroxychloroquine, cyclophosphamide, thalidomide, and/or infliximab
* Patients able to provide written consent

Exclusion Criteria:

* Patients on pulmonary vasodilator drugs (flolan, remodulin, bosentan, sildenafil) n the prior 28 days. Patients on stable dose of calcium channel blocker for more than 1 month prior to right heart catheterization can be continued on the calcium channel blocker.
* Patients with severe airway obstruction as defined by FEV1/FVC of less than 35%
* Patients with World Health Organization (WHO) class IV status.
* Patients who are pregnant or breast feeding
* Patients with significant left ventricular dysfunction with a left ventricular ejection fraction of less than 35%
* Cardiac index < 2.0 liters and/or right atrial pressure >15 mm Hg
* Significant liver dysfunction not due to sarcoidosis.
* Patients with severe other organ disease felt by investigators to impact on survival during the course of the study.
* Patients unable to perform the 6 minute walk study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-04; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in six minute walk distance | 16 weeks

SECONDARY OUTCOMES:
Change in pulmonary hemodynamics | 16 weeks
Improvement in quality of life with therapy | 48 weeks
Safety of treatment | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (4):
- United States (4):
  - Mount Sinai, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Baughman RP, Culver DA, Cordova FC, Padilla M, Gibson KF, Lower EE, Engel PJ. Bosentan for sarcoidosis-associated pulmonary hypertension: a double-blind placebo controlled randomized trial. Chest. 2014 Apr;145(4):810-817. doi: 10.1378/chest.13-1766. PMID 24177203